CLINICAL TRIAL: NCT01541696
Title: Exchangeable Zn Pool Size and Zn Absorption From Sprinkles and Traditional Foods in Pakistani Infants/Toddlers
Brief Title: Exchangeable Zinc Pool Size and Zn Absorption From Sprinkles and Traditional Foods in Pakistani Infants /Toddlers
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: University of Colorado, Denver (Other); International Atomic Energy Agency (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Shabina Ariff, Assistant Professor, Aga Khan University
Other Study IDs: 1387-PED-ERC-09
Record Dates: First submitted 2012-01-11; First posted 2012-03-01 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Malnutrition
Keywords: zinc; zn; EZP (exchangeable zinc pools)multivitamin MN
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group B: subjects in this group will receive Micronutrient Supplements only.
- Group C: Subjects in this Group will receive Micronutrient Supplements plus Zinc.

SUMMARY:
The broad objective is to improve zinc status in older infants and young children who are at risk of zinc deficiency because of combination of inadequate dietary zinc intake and high rates of diarrhea. As a sub-study within larger RCT using zinc fortified Sprinkles, the proposed study will measure the amount of zinc absorbed from a test meal of typical unfortified complementary foods consumed by Pakistani infants, or the same complementary foods fortified by the addition of the Zn-containing Sprinkle.

DETAILED DESCRIPTION:
In the nested study we aim to measure from a subgroup of recruited children in the main study, the amount of zinc absorbed from typical unfortified complementary foods consumed by Pakistani infants, and compare it with the same complementary food fortified by the addition of the Zn-containing Sprinkles and multi vitamins. Since EZP Exchangeable Zinc Pool is considered to be the gold standard for estimation of the actual concentration of zinc in the plasma that is readily available for cellular function, we would also calculate the EZP in this subset of samples.

The specific aim of the nested study will :

1. Determine absorption of zinc (Zn) from a test meal consisting of typical local food with addition of a multiple-micronutrient Sprinkles product containing (10 mg of Zn) vs absorption from the same meal without zinc supplementation to those with no micronutrient fortification.
2. Compare size of exchangeable Zn pool (EZP) for subjects who have been randomized to receive multi-micronutrient Sprinkle (MN) only with those who were randomized to (MN+Zn ) with control group.
3. Children will be followed for growth monitoring for at least 2 years.
4. Plasma zinc and phytates levels in the weaning diet will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Infants between the ages of 9 and 12 months and on weaning diet for at least 3 months.
* Infants who are currently recruited in the main zinc gates study and consuming sprinkles sachet containing micronutrient and zinc .

Exclusion Criteria:

* Infants with congenital anomalies
* Infants not on weaning diet
* Infants not consuming sprinkles sachet containing micronutrients

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants between the ages of 9 and 12 months
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Exchangeable Zn Pool Size and Zn Absorption from Sprinkles and Traditional Foods in Pakistani Infants/Toddlers | one year
  Compare size of exchangeable Zn pool (EZP) for subjects who have been randomized to receive multi-micronutrient Sprinkle (MN) only with those who were randomized to (MN+Zn ) .
  Compare plasma zinc levels between the two groups Measure the fractional absorption of zinc between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, MBBS, FCPS, Principal Investigator — Aga Khan University; Shabina Ariff, MBBS, FCPS, Study Director — Aga Khan University; Zulfiqar A Bhutta, PhD, Study Chair — Aga Khan University
Locations (1):
- Bilal Colony, Karachi, Sindh, Pakistan